CLINICAL TRIAL: NCT01056302
Title: Advanced Visuohaptic Surgical Planning for Trauma Surgery
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: F7124-R
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Maxillofacial Injuries
Keywords: Reconstructive surgical procedures; visuohaptic
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: 15 patients who underwent surgical repair of mandibular fractures at San Francisco VA Medical Center
  Interventions: Procedure: Surgical repair of mandibular fractures

INTERVENTIONS:
Procedure: Surgical repair of mandibular fractures — Patients will undergo whatever needed surgical repair of maxillofacial trauma that is necessary. Records such as CT imaging and plaster models of the jaws will be utilized in the standard way to plan and carry out the surgery. The CT scan will also be used within the visuohaptic computational environment to develop and evaluate the user interface. The amount of time taken to work up and plan surgery using standard surgical practice and using the computational platform will be compared. Real surgical outcome will be compared to the simulated surgical outcome using the proposed software tool.

SUMMARY:
This study proposes to develop a computer-based software tool that will allow surgeons to plan and simulate surgery for patients with jaw trauma.

DETAILED DESCRIPTION:
The proposed tool will allow surgeons from different specialties to simulate, plan and iterate on complex procedures based on individual patient data in 3-D from a CT scan. The software will allow surgeons to both see and feel the results of their interventions - for example, the quality of the bite or bone alignment of a reconstructed jaw following severe trauma - before the actual surgery, leading to better planning, fewer errors, shortened surgery time and improved outcomes for the patients. The purpose of this study is the evaluation of a visuohaptic planning system for mandibular trauma surgery that is based on interactive manipulation of CT data.

ELIGIBILITY:
Inclusion Criteria:

* Craniofacial deformity, including post-traumatic, congenital or acquired deformity
* Patients who have already have surgery because there was a clinical indication for surgical correction

Exclusion Criteria:

* No craniofacial deformity
* No clinical indication for surgical correction
* Contraindication for surgical correction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will veterans who present to the Oral/Maxillofacial Surgery Clinic at the San Francisco VA Medical Center. The study will use pre-existing data from patients undergoing reconstructive facial surgery at the San Francisco VA with clinic indications that require preoperative CT scans and preoperative radiographs as well as model casts.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebeka Silva, DMD, Principal Investigator — VA Medical Center, San Francisco
Locations (1):
- VA Medical Center, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schvartzman SC, Silva R, Salisbury K, Gaudilliere D, Girod S. Computer-aided trauma simulation system with haptic feedback is easy and fast for oral-maxillofacial surgeons to learn and use. J Oral Maxillofac Surg. 2014 Oct;72(10):1984-93. doi: 10.1016/j.joms.2014.05.007. Epub 2014 May 24. PMID 25234531
- [Result] Forsslund J, Chan S, Selesnick J, Salisbury K, Silva RG, Blevins NH. The effect of haptic degrees of freedom on task performance in virtual surgical environments. Stud Health Technol Inform. 2013;184:129-35. PMID 23400144
- [Result] Girod S, Schvartzman SC, Gaudilliere D, Salisbury K, Silva R. Haptic feedback improves surgeons' user experience and fracture reduction in facial trauma simulation. J Rehabil Res Dev. 2016;53(5):561-570. doi: 10.1682/JRRD.2015.03.0043. PMID 27898160

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: 3 patients with maxillofacial trauma who underwent surgical repair at San Francisco VA Medical Center
  Surgical repair of maxillofacial trauma: Patients will undergo whatever needed surgical repair of maxillofacial trauma that is necessary. Records such as CT imaging and plaster models of the jaws will be utilized in the standard way to plan and carry out the surgery. The CT scan will also be used within the visuohaptic computational environment to develop and evaluate the user interface. The amount of time taken to work up and plan surgery using standard surgical practice and using the computational platform will be compared. Real surgical outcome will be compared to the simulated outcome using the proposed software tool.
Period: Overall Study
Arm/Group | Group 1
Started | 3
Completed | 3 (The study was completed with 3 datasets from patients who had maxillofacial trauma and were treated)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Patients who underwent mandibular fracture repair had their age documented in the medical record.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 60 [58 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3
Presence of mandibular fracture [Number; unit: fractures] — The number of mandibular fractures for all participating patients was recorded. Each patient underwent a preoperative workup, including CT scan, to count the number of fractures present within the mandible.
  fractures
    Number of total fractures | 5
    Number of condylar fractures | 2
    Number of angle fractures | 3
Degree of mandibular fracture displacement [Number; unit: Fractures] — The mandibular fractures for all participating patients were described in terms of degree of displacement using standard medical terminology (nondisplaced, mild-, moderate- or severely displaced). Each patient underwent a preoperative workup, including clinical examination and CT scan, in order to assess the degree of fracture displacement.
  Fractures
    Non-displaced fracture | 0
    Mildly displaced fracture | 0
    Moderately displaced fracture | 2
    Severely displaced fracture | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Deviation From Actual Surgical Outcome During Virtual Repair of Mandibular Fractures, Using the Novel Visuohaptic Computational Platform That Was Developed by the Investigators
Description: The virtual surgical outcome was compared to the actual surgical outcome. This was accomplished by measuring distances (mm) and angles between specific mandibular anatomic points in the virtual environment and comparing it to the same distances (mm) and angles between specific mandibular anatomic points in the actual surgical outcome, as seen in a 3D rendering derived from the patient's postoperative CT scan. The actual surgical repair was considered to be the gold standard. A deviation of more than 10% between the virtual surgical repair and the actual surgical repair was considered to be above threshold (inaccurate virtual fracture repair).
Time Frame: 6 months
Population: All participants were diagnosed with acute mandibular fracture(s) and underwent surgical repair of the fracture(s) at the San Francisco VA Medical Center
Measure: Mean (95% Confidence Interval); unit: percentage of measurement deviation
Groups:
- Group 1: 3 patients with mandibular fracture(s) who underwent surgical repair at San Francisco VA Medical Center
  Patients underwent surgical repair of their mandibular fracture(s) in the usual and customary way. Preoperative CT imaging was utilized by the surgeon to plan and carry out the surgery. Following surgery, a postoperative CT scan was done to assess the success of the surgery to accurately reposition all the fractured bone. Each patient's preoperative CT scan was also used within the visuohaptic computational environment to develop and evaluate the user interface. Once the software was deemed suitable for use, it was tested. The test consisted of measuring the accuracy of the virtual surgical repair compared to the real surgical outcome, as seen on the postoperative CT scan.
Arm/Group | Group 1
Number analyzed (Participants) | 3
percentage of measurement deviation | 5 [1 to 7]

2. Secondary Outcome: Development and Evaluation of Automation Features for the Visuohaptic Virtual Surgery Planning Environment
Description: The addition of automation features for the visuohaptic virtual surgical planning environment was envisioned to make it possible to predict the number, type, size, and position of reconstruction hardware (bone plates and screws) that would best fit the virtually repaired mandibular fractures. The goal was to compare the hardware configuration selected and used in the actual surgical repair for the 3 participating patients with what the software predicted. Unfortunately, the software development proved to be difficult to add this automated feature.
Time Frame: 3 years
Population: The automation feature was envisioned to predict size and position of bone plates/screws that would best fit the virtually repaired mandibular fractures. The goal was to compare the actual hardware configuration with what the software predicted. The software development proved too difficult to add this automated feature. Data were not collected.
Groups:
- Group 1: Patients with mandibular fracture(s) who underwent surgical repair at San Francisco VA Medical Center
  Patients underwent surgical repair of their mandibular fracture(s) in the usual and customary way. Preoperative CT imaging was utilized by the surgeon to plan and carry out the surgery. Following surgery, a postoperative CT scan was done to assess the success of the surgery to accurately reposition all the fractured bone. Each patient's preoperative CT scan was also used within the visuohaptic computational environment to develop and evaluate the user interface. Once the software was deemed suitable for use, it was tested. The test consisted of measuring the accuracy of the virtual surgical repair compared to the real surgical outcome, as seen on the postoperative CT scan.
Arm/Group | Group 1
Number analyzed (Participants) | 0

3. Secondary Outcome: Implementation and Test of the Telemedicine Prototype
Description: Measurement of the accuracy of the virtual surgical repair generated by the surgeon operating the software when a remote surgeon digitally sends a CT scan of a patient with an acute mandibular fracture(s). The telemedicine interface would require an automated method to segment the CT scan into the fractured components. The operator would manipulate the bone fractures, select the hardware type and size for "best fit", and generate a report back to the remote surgeon.
Time Frame: 3 years
Population: The telemedicine prototype, which would allow an operator to quickly create a virtual surgical plan to send to a remote surgeon, predicting needed reconstructive hardware, could not be developed due to software limitations. Data were not collected.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Group 1: 3 patients with mandibular fracture(s) who underwent surgical repair at San Francisco VA Medical Center
  Surgical repair of mandibular fracture(s): Patients will undergo whatever needed surgical repair of mandibular fracture(s) that is necessary. Records such as CT imaging were utilized in the standard way to plan and carry out the surgery. The CT scan was also used within the visuohaptic computational environment to develop and evaluate the user interface.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes